CLINICAL TRIAL: NCT02454816
Title: Introduction Study of Dual HIV & Syphilis Rapid Diagnostic Tests in Antenatal Clinics in COLOMBIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HIV2.0
Record Dates: First submitted 2015-05-12; First posted 2015-05-27 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Syphilis; HIV
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Intervention Model Description: A cluster randomised controlled trial will be conducted in 12 health facilities (4 hospitals and 8 health centres) in Bogota and Cali, Colombia.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single HIV RDT and single syphilis RDT (Experimental): It is a diagnostic intervention, at the cluster level This arm includes a single (separate) rapid test for HIV and Syphilis. In this case pregnant women enrolled are sampled with two drops of blood (one for each cassette). Positive patients for syphilis are treated immediately and reactive patients for HIV continue with their diagnostic algorithm, in any case patients receive appropriate counseling
  Interventions: Device: Single HIV RDT and single syphilis RDT
- Dual HIV/syphilis RDT (Active Comparator): It is a diagnostic intervention, at the cluster level. This arm includes a dual rapid test for HIV and syphilis, which means that in the same cassette will be available the information about the results for both conditions. In this case pregnant women enrolled are sampled with one drop for the cassette, which is enough to get both of the results. Positive patients for syphilis are treated immediately and reactive patients for HIV continue with their diagnostic algorithm, in any case patients receive appropriate counseling
  Interventions: Device: Dual HIV/syphilis RDT

INTERVENTIONS:
Device: Single HIV RDT and single syphilis RDT — It is a diagnostic intervention, at the cluster level This arm includes a single (separate) rapid test for HIV and Syphilis. In this case pregnant women enrolled are sampled with two drops of blood (one for each cassette). Positive patients for syphilis are treated immediately and reactive patients for HIV continue with their diagnostic algorithm, in any case patients receive appropriate counseling
  Arms: Single HIV RDT and single syphilis RDT
Device: Dual HIV/syphilis RDT — It is a diagnostic intervention, at the cluster level. This arm includes a dual rapid test for HIV and syphilis, which means that in the same cassette will be available the information about the results for both conditions. In this case pregnant women enrolled are sampled with one drop for the cassette, which is enough to get both of the results. Positive patients for syphilis are treated immediately and reactive patients for HIV continue with their diagnostic algorithm, in any case patients receive appropriate counseling
  Arms: Dual HIV/syphilis RDT

SUMMARY:
Global and regional initiatives have been launched for the dual elimination of mother-to-child transmission (MTCT) of HIV and syphilis. As one of the important components in the initiatives, early detection and timely intervention of pregnant women infected with HIV and/or syphilis is critical. In order to improve the number of women tested and treated, innovative strategies are needed.

Serologic tests are the diagnostic tests of choice for HIV and syphilis. There are two types of serological tests (treponemal and non-treponemal tests) for diagnosis of syphilis. These generally require venous blood for screening of symptomatic and asymptomatic patients. In addition, these tests are technically demanding, and require laboratory equipment which is not widely available in most resource-limited settings.

Recently, Rapid diagnostic tests (RDTs) that can be used at point-of-care for simultaneously detecting antibodies to HIV and syphilis (dual HIV & syphilis treponemalRDTs) using serum/plasma, venous whole blood, or finger-stick whole blood have been developed and are now commercially available.

In low-resource settings, a combination of two or three rapid diagnostic tests (RDTs), in which one screening test with a second test to confirm initial positive results or two RDTs in parallel with a third test as a tiebreaker for discordant samples, can be used to diagnose HIV on finger-stick blood. To date, there are few data on the implications of using these RDTs in the antenatal clinic settings, although they have been evaluated in laboratory-based studies and shown encouraging sensitivities and specificities as compared with reference laboratory tests.

The objective of this research is to assess the uptake of syphilis testing after the introduction of dual HIV/syphilis rapid testing as compared to single rapid syphilis testing in antenatal clinics in Colombia.

The secondary objectives of the study are: To determine the uptake of treatment of syphilis after the intervention, To determine the uptake of HIV testing in ANC attendees after the intervention, To explore the acceptability of dual HIV/syphilis RDTs by ANC attendees and health workers, To assess the organizational and socio-cultural advantages and barriers to introduction with a aim of sustainable adoption of dual HIV/syphilis RDTs in antenatal services, To determine the workload and cost implications of introduction of dual HIV/syphilis RDTs in antenatal services

DETAILED DESCRIPTION:
Methods:

Desing: Cluster randomized trial including and quantitative component, a qualitative component (in-deep interviews)and a time and cost estimation component in the antenatal care setting.

Population: Primary health facilities (n=12) in Bogotá and Cali, Colombia. Eligibility criteria: Inclusion Criteria: Pregnant women attending first ANC visit at the study sites, or women not previously tested in this pregnancy,Women aged 14 years old or above, Any woman who has tested positive for HIV and/or syphilis in the past (will be permitted to enrol), Women providing a written informed consent.Exclusion Criteria: Women who have already been enrolled in this study, Women < 14 years of age, Women unable to provide informed consent.

Test to be evaluated: Each of the 12 institutions participating in the trial were assigned in a random way to rapid single test for HIV and Syphilis or dual rapid test HIV/syphilis. The brand of the rapid test selected for the study, passed throw a process of selection by the National Health Institute in Colombia, in order to choose the best test according to desirable performance and operational characteristics. The brand Standard Diagnostics the Bioline was donated to do the rapid test in the present study with pregnant women.

Analysis:

* CONSORT diagram for the cluster randomized trial will be shown.
* Primary analysis will be based on intention-to-treat principle, with no facility excluded from analysis after the random assignment.
* Baseline characteristics of clusters (facilities) and of the women enrolled in each arm will be provided.
* For qualitative variables frequencies and percentages will be reported. For quantitative normally distributed variables, the number of subjects, means and standard errors will be provided, while medians, interquartile range, minima and maxima will be reported for skewed non-normal quantitative variables.
* Because of the clustered nature of outcomes due to randomization to interventions based on clusters (facilities), the Generalized Estimating Equations (GEE) modelling, with binomial distribution and logit link, will be used to estimate the risk difference (RD) and odds ratio (OR) of Syphilis testing, Syphilis treatment and HIV testing uptake, with 95% Confidence Interval, adjusted for clustering, between interventions arms A and B. This model will adjust for any important baseline factors, including whether any testing in Syphilis or HIV was ever done previously.
* Intra-cluster correlations (ICC) for overall, as well as ICCs stratified for important baseline factors of interest, will be estimated.
* Two-sided tests and 5% significance levels will be used, and 95% confidence intervals for all relevant parameters. SAS statistical packages will be used for the statistical analyses.

Expected results: The results of the study will be used in the design of strategies of policies/national o local guidelines or even screening antenatal programs for HIV and syphilis, the development of the best practice to the adoption of the rapid test for HIV and Syphilis. The information collected will be used to share the experience and the lessons learned to other countries in order to development guidelines of global, regional and national policies to implement in order to impact the transmission of maternal-child HIV and syphilis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending first ANC visit at the study sites, or women not previously tested in this pregnancy
* Women aged 14 years old or above
* Any woman who has tested positive for HIV and/or syphilis in the past (will be permitted to enrol)
* Women providing a written informed consent

Exclusion Criteria:

* Women who have already been enrolled in this study
* Women < 14 years of age
* Women unable to provide informed consent

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants in syphilis testing with SRDT compared to DRDT post intervention | 4 months

SECONDARY OUTCOMES:
Differences in Number of participants with uptake of HIV testing between Arm A and Arm B. | 4 months
Number of participants with syphilis treatment between Arm A and Arm B | 4 months
Number of participants with uptake of syphilis treatment between Arm A and Arm B | 4 months
Number of participants with acceptability and feasibility of dual RDTand health care workers. | 4 months
Determine the workload and cost implications of the introduction of dual RDTs in antenatal services through a time/motion/cost exercise. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Carlos Holmes Trujillo, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Obure CD, Gaitan-Duarte H, Losada Saenz R, Gonzalez L, Angel-Muller E, Laverty M, Perez F. A comparative analysis of costs of single and dual rapid HIV and syphilis diagnostics: results from a randomised controlled trial in Colombia. Sex Transm Infect. 2017 Nov;93(7):482-486. doi: 10.1136/sextrans-2016-052961. Epub 2017 May 11. PMID 28495681